CLINICAL TRIAL: NCT01283529
Title: Reference Values for Cardiac Output and Blood Volume Variables in Children With Normal Cardiac Function Measured Under General Anesthesia.
Brief Title: Reference Values for Pulse Induced Continuous Cardiac Output (PiCCO) Variables in Children
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Gunnar Bentsen, Consultant, Oslo University Hospital
Other Study IDs: 2010/27693; 2010/2576-4 (Other: Ethics commitee)
Record Dates: First submitted 2011-01-17; First posted 2011-01-26 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Reference Values
Keywords: Intrathoracal blood volume; Cardiac output; Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children 0 - 15 years: Children undergoing neurosurgery in general anesthesia

SUMMARY:
Pulse induced continuous cardiac output (PiCCO) is an established technology for measurement of advanced hemodynamic variables in critically ill patients. PiCCO is approved and designed also for use in children, but there is a lack of documentation of reference values in children not suffering from a critical illness. The goal of this study is to establish such values.

ELIGIBILITY:
Inclusion Criteria:

* Age < 15 years
* Scheduled for major neurosurgery in general anesthesia

Exclusion Criteria:

* Cardiac disease
* Infection / sepsis

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 40 children age 0 - 15 years undergoing major neurosurgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-01; Primary Completion 2014-02 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Reference values for PiCCO variables | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Bentsen, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Oslo County, Norway